CLINICAL TRIAL: NCT00432874
Title: A Prospective Evaluation of the Safety and Efficacy of Two Forms of Corneal Stromal Hydration
Brief Title: Prospective Evaluation of Safety and Efficacy of Two Forms of Corneal Stromal Hydration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Dr. Mark Mifflin, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: UT16122
Record Dates: First submitted 2007-02-06; First posted 2007-02-08 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-10

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Anterior stromal hydration ("Wong" method)
  Interventions: Procedure: wound hydration method
- 2 (Active Comparator): Traditional lateral wound hydration
  Interventions: Procedure: wound hydration method

INTERVENTIONS:
Procedure: wound hydration method — Anterior vs lateral wound hydration

SUMMARY:
The study objective is to compare traditional and Wong methods of wound hydration for wound sealing following cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Visually significant cataract requiring surgery

Exclusion Criteria:

* Evidence of Fuch's dystrophy, anterior basement membrane dystrophy, or corneal thinning or scarring
* Any intraoperative complications
* Cataract incision length < 1 mm
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-02; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Proportion of eyes with wound leakage at the end of surgery | Intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Mifflin, MD, Principal Investigator — University of Utah
Locations (1):
- John Moran Eye Center, Salt Lake City, Utah, United States